CLINICAL TRIAL: NCT03897673
Title: Optimizing Benefits While Reducing Risks of Iron in Malaria-endemic Areas
Acronym: OptiM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: STUDY00001235
Record Dates: First submitted 2019-03-28; First posted 2019-04-01 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Iron Deficiency Anemia; Iron-deficiency; Anemia, Iron Deficiency; Anemia; Anemia in Children; Malaria
MeSH Terms: conditions — Anemia, Iron-Deficiency; Anemia; Malaria

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Early Iron (Experimental): Children in the immediate iron group will receive iron syrup for the first three months (84 days) and placebo syrup for the fourth month.
  Interventions: Dietary Supplement: Early Iron
- Delayed Iron (Experimental): Children in the delayed iron group will receive placebo syrup for the first month (28 days) and iron syrup for the second, third, and fourth months.
  Interventions: Dietary Supplement: Delayed Iron
- Community Control Children (No Intervention): Healthy, non-anemic community children will be enrolled from the same households and villages as the children with malaria. They will not have ZPP tested or receive iron, but they will also be under the same illness surveillance as the children with malaria.

INTERVENTIONS:
Dietary Supplement: Early Iron — iron syrup for the first three months (84 days) and placebo syrup for the fourth month
  Arms: Early Iron
Dietary Supplement: Delayed Iron — placebo syrup for the first month (28 days) and iron syrup for the second, third, and fourth months
  Arms: Delayed Iron

SUMMARY:
Daily iron (ferrous sulfate, 2 mg/kg/day) or placebo syrup for first four months (112 days) of the 12-month (336-day) study. Children in the immediate iron group will receive iron syrup for the first three months (84 days) and placebo syrup for the fourth month. Children in the delayed iron group will receive placebo syrup for the first month (28 days) and iron syrup for the second, third, and fourth months.

DETAILED DESCRIPTION:
Provision of sufficient iron for brain development in children living in malaria-endemic areas while also protecting them from infection is an unachieved public health goal for >10 years. The 2006 landmark study on malaria-endemic Pemba Island brought the complicated relationship between iron and malaria to the world stage by reporting universal prophylactic iron supplementation increases the risk of child hospitalization and death. Treating iron deficiency in children who have malaria is also an unsolved challenge. In sub-Saharan Africa, iron deficiency and malaria coexist, frequently causing a multifactorial anemia that is a primary cause of hospitalization and mortality in children <5 y. The current World Health Organization standard-of-care regimen of concurrent treatment with antimalarial medication and iron therapy has been unsuccessful, with frequent reports of subsequent infection, including malaria, persistent iron deficiency, and unresolved anemia.

One solution to effectively treat coexisting malaria and iron deficiency is to stagger interventions, treating malaria first and delaying iron. The inflammatory response against malaria induces high levels of the protein hepcidin, which reduces intestinal iron absorption and prohibits release of iron from reticulo-endothelial cells. Iron given orally during or shortly after a malaria episode is thus not well absorbed or distributed to red blood cells or the brain. Moreover, unabsorbed iron in the gut may promote the growth of pathogenic bacteria, potentially leading to subsequent infectious morbidity. A pilot study was recently completed in Ugandan children with malaria and iron deficiency that used iron stable isotopes to test whether iron given 28 days after (delayed group) or concurrently with (immediate group) antimalarial treatment was better incorporated into red blood cells (1R03HD074262). It was found that delayed iron was incorporated twice as well as immediate iron and that iron status at 56 days was similar between groups. An important finding was that children in the immediate group had a higher incidence of infections in the 56-day follow-up period. In this application, the team proposes a large-scale, randomized clinical trial with 12 months follow up powered to capture long-term differences in iron status, morbidity, and neurobehavioral development as a function of immediate or delayed iron following treatment for malaria and iron deficiency. The gut microbiome will be analyzed to elucidate a mechanism of any differences in incidence of infections.

One long-term goal is to develop safe and effective strategies for managing concurrent malaria and iron deficiency in children, with reduction of infections and optimization of neurobehavioral development representing successful outcomes. The objective of this application is to conduct a placebo-controlled, randomized clinical trial to determine whether iron therapy begun with vs. 28 days after antimalarial treatment in Ugandan children 6-48 months with malaria and iron deficiency leads to better iron status, fewer infections, and better neurobehavioral development after 12 months. The central hypothesis is that better iron incorporation and lower incidence of infectious illness observed with delayed iron in our short-term, physiology-focused R03 study will translate into better long-term iron status, fewer episodes of infection, and better neurobehavioral outcomes after 12 months. The rationale is that this study will determine if staggering antimalarial treatment and iron therapy protects against immediate morbidity while also optimizing long-term neurobehavioral development. The Specific Aims are:

Aim 1: Establish the effect of immediate vs. delayed iron treatment on long-term iron status.

It is hypothesized that delayed iron will result in better iron status 6 and 12 months after treatment for malaria due to better initial iron absorption and utilization as compared to the immediate iron group.

Aim 2: Determine the effect of delayed iron treatment on the incidence of infectious illness.

It is hypothesized that the better absorbed delayed iron will result in fewer infections in the 6 and 12 months after treatment for malaria due, in part, to a less pathogenic intestinal microbiome profile.

Aim 3: Establish the effect of delayed iron treatment on neurobehavioral development.

It is hypothesized that delayed iron will result in better neurobehavioral outcomes (as assessed by standardized cognitive and behavioral tests) due to better iron absorption and utilization.

Anticipated Impact: Untreated iron deficiency may protect a child from malaria and other infections, but the consequent potentially permanent damage to the developing brain is an unacceptable alternative. Establishment of methods to effectively ensure brain iron health while protecting the child from infection will promote attainment of full cognitive and behavioral development for tens of millions of children worldwide suffering from malaria and iron deficiency.

ELIGIBILITY:
Inclusion Criteria for children with malaria:

* Hemoglobin 7.0 - 9.9 g/dL
* ZPP > = 80 µmol/mol heme
* P. falciparum positive by Giemsa smear or RDT positive
* Temperature ≥ 37.5C or history of fever in past 24 hours

Exclusion Criteria for Children with Malaria:

* Any WHO criterion for severe malaria, including severe anemia, prostration, cerebral malaria, repeated seizures or symptoms like persistent vomiting, high temperature (>39.5°C), or tea-colored urine
* Severe malnutrition, as evidenced by severe wasting or bilateral pitting edema
* Known sickle cell disease
* Acute hemorrhage
* Known cancer or leukemia
* Caregiver does not understand English or Luganda

Inclusion Criteria for Community Children:

* Same neighborhood, extended household or nearby neighborhood of a child with malaria
* Same age group as a child with malaria
* Hemoglobin > = 10.0 g/dL

Exclusion Criteria for Community Children

* Clinical malaria infection or any active illness within the past 4 weeks requiring medical care
* Chronic illness requiring medical care
* Major medical abnormalities on screening history or physical exam, including measured temperature ≥ 37.5°C
* Known developmental delay or neurologic disorder
* Prior history of coma
* Caregiver does not understand English or Luganda
* Other severe illness such as pneumonia or cardiac failure

Ages: 6 Months to 48 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 600 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Prevalence of iron deficiency | 6-months
  Number of participants who are iron deficient (defined as a zinc protoporphyrin (ZPP) concentration greater than or equal to 80 umol/mol heme) at 6-months follow-up in the early iron vs. delayed iron treatment groups
All-cause incidence of infectious illness | 6-months
  Number of participants who report an infection and total number of infections reported to a study medical officer in the early iron vs. delayed iron treatment groups. This includes all infectious illness including clinical malaria episodes.
Effect on neurobehavioral development: BRS | 12-months
  Behavior Rating Scales (BRS) scores at 12 months follow up in the early iron vs. delayed iron treatment groups. BRS assesses socioemotional behavior. Scores range from 1-5. Higher raw scores for Fearful/Wary Affect, Negative Affect, and Hyperactivity/Over-activity indicate less optimal behavior, as do lower raw scores for Positive Affect, Adaptation to Change, Exploration and Activity Level.
Effect on neurobehavioral development: MSEL | 12-months
  Mullen Scales of Early Learning (MSEL) scores at 12 months follow up in the early iron vs. delayed iron treatment groups.The MSEL assesses motor, visual, and language ability and is used to measure cognitive ability. Scores from fine motor, visual reception, receptive language, and expressive language scales are summed to give the early learning composite score, a measure of overall cognitive ability. Each sub-scale is standardized to calculate a standard score, percentile, and age-equivalent score. Composite scores range from 0 to 100 with 100 indicating greater cognitive ability.

SECONDARY OUTCOMES:
ZPP | 12-months
  Prevalence of zinc protoporphyrin (ZPP) ≥ 80 umol/mol heme in the early iron vs. delayed iron treatment groups
Iron status: Hemoglobin | 6- and 12-months
  Concentrations of hemoglobin in the immediate vs. delayed groups
Iron status: ferritin | 6- and 12-months
  Concentrations of ferritin in the early iron vs. delayed iron treatment groups
Iron status: soluble transferrin receptor (sTFR) | 6- and 12-months
  Concentrations of sTFR in the early iron vs. delayed iron treatment groups
Iron status: hepcidin | 6- and 12-months
  Concentrations of hepcidin in the early iron vs. delayed iron treatment groups
Iron status: C-reactive Protein (CRP) | 6- and 12-months
  Concentrations of CRP in the early iron vs. delayed iron treatment groups
All-cause infectious episodes | 12-months
  Incidence of all-cause infectious episodes and incidence of clinical malaria episodes during the 12-months follow-up period; incidence of all-cause and malaria-specific hospitalizations
Proteobacteria | Baseline, 6-months, 12-months
  Change in relative fecal abundance of Proteobacteria
Child Behavior Checklist (CBCL) | 12-months
  CBCL scores at 12 months follow up. Preschool Child Behavioral Checklist (P-CBCL) is a parent-report checklist that assesses internalizing, externalizing, and total behavioral problems. Higher scores indicate more problematic behavior or diminished function.
Behaviors Related to Executive Function (BRIEF) | 12-months
  BRIEF scores at 12 months follow up. Behavior Rating Inventory of Executive Functioning, Preschool edition (BRIEF-P) is a parent-report checklist that assesses global executive function. Higher scores indicate more problematic behavior or diminished function.

CONTACTS AND LOCATIONS:
Locations (1):
- Kampala, Uganda, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No